CLINICAL TRIAL: NCT07388056
Title: Efficacy and Safety of Extended Anticoagulant Therapy in Cancer Associated Thrombosis-A Ten Year Retrospective Study.
Brief Title: Efficacy and Safety of Extended Anticoagulant Therapy in Cancer Associated Thrombosis in Thai Population
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Lantarima Bhoopat, Hematology, Internal medicine, Faculty of medicine, Thammasat University
Other Study IDs: MTU-EC-IM-1-301/65
Record Dates: First submitted 2026-01-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cancer-associated Thrombosis
MeSH Terms: interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Therapeutic dose anticoagulant group: including patients with the standard therapeutic dose-administered after the initial six-month treatment period.
  Interventions: Drug: Anticoagulant
- Prophylactic dose anticoagulant group: including patients with the doses lower than therapeutic dose-administered at any point after the initial six-month treatment period.
  Interventions: Drug: Anticoagulant

INTERVENTIONS:
Drug: Anticoagulant — warfarin at therapeutic level (INR 2-3), Low molecular weight heparin (LMWH) DOAC

SUMMARY:
The goal of this observational study is to learn about the long-term efficacy and safety of extended anticoagulant treatment in patients with cancer associated thrombosis. (CAT) The main question it aims to answer is:

• Does extended prophylactic dose anticoagulant provide comparable efficacy and safety to therapeutic dosing after 6-month treatment of anticoagulant? The medical record data of participants who's already received for at least 6-month anticoagulant treatment upon regular medical care for CAT will be collected and analyzed about their recurrent thrombosis, anticoagulant related bleeding, and survival outcome.

DETAILED DESCRIPTION:
Adult patients aged ≥18 years with histopathological confirmed cancer, treated at Thammasat University Hospital and Panyananthaphikkhu Chonprathan Medical Center between January 2012 and December 2022, were eligible for inclusion.

Patients were initially screened using ICD-10 diagnostic codes C00-D009 for malignancy in conjunction with codes for venous thromboembolism (I82.-, other venous embolism and thrombosis; K55.0, mesenteric vein thrombosis; I82.0, hepatic vein thrombosis; K75.1, phlebitis of the portal vein; and I26.-, pulmonary embolism). Eligible patients required to have a radiologically confirmed diagnosis of cancer-associated thrombosis (CAT) and to have received anticoagulation therapy for at least six months. Clinical data were extracted from the Computerized Provider Order Entry (CPOE) system.

ELIGIBILITY:
Here's a polished version of your Inclusion and Exclusion Criteria section with grammar, spelling, and phrasing corrected for clarity and formal research style:

Inclusion Criteria

* Adult patients aged ≥18 years
* Histopathologically confirmed cancer
* Radiologically confirmed diagnosis of cancer-associated thrombosis (CAT)
* Received anticoagulation therapy for at least six months Exclusion Criteria
* Patients who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at Thammasat University Hospital or Panyananthaphikkhu Chonprathan Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrent thrombosis | After completing 6-month of treatment to the time that anticoagulant stop or recurrent thrombosis occurred through study completion, at the end of December 2025.
  cumulative incidence of recurrent thrombosis

SECONDARY OUTCOMES:
Anticoagulant related bleeding | After completing 6-month of treatment to the time that anticoagulant stop or bleeding occurred through study completion, at the end of December 2025.
  cumulative incidence of bleeding
Overall survival | The time from VTE diagnosis to last follow up or die through study completion, at the end of December 2025.
  Overall survival

IPD SHARING:
Plan to Share IPD: Undecided